CLINICAL TRIAL: NCT00002563
Title: Health Status and Quality of Life in Patients With Early Stage Hodgkin's Disease: A Companion Study to SWOG-9133
Brief Title: SWOG-9208 Quality of Life and Health Status in Patients With Stage I or Stage II Hodgkin's Disease
Status: Completed | Type: Observational
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Cancer and Leukemia Group B (Network)
Responsible Party: Sponsor
Other Study IDs: CDR0000063515; U10CA032102 (NIH); SWOG-9208 (Other: SWOG); CLB-9497 (Other: CALGB)
Record Dates: First submitted 1999-11-01; First posted 2004-07-19 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Lymphoma; Psychosocial Effects of Cancer and Its Treatment
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; psychosocial effects of cancer and its treatment
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Psychiatric Rehabilitation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: psychosocial assessment and care — Evaluate psychosocial function at prestudy, 6 months after starting treatment on S9133, and annually at 1-7 years after starting treatment on S9133.
Procedure: quality-of-life assessment — Evaluate quality of life at prestudy, 6 months after starting treatment on S9133, and annually at 1-7 years after starting treatment on S9133.

SUMMARY:
RATIONALE: Quality-of-life assessment in patients undergoing cancer treatment may help determine the intermediate- and long-term effects of treatment on patients with cancer.

PURPOSE: This clinical trial studies the impact of therapy on the health status and quality of life of patients with stage I or stage II Hodgkin's disease who are receiving radiation therapy with or without chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate prospectively the health status and quality of life of patients with Stage I/IIA Hodgkin's disease randomized on protocol SWOG-9133 (CLB-9391) to treatment with subtotal nodal irradiation with vs. without 3 courses of doxorubicin/vinblastine. II. Describe the short-term effects of these treatments on these patients and compare their impact on quality of life (i.e., patient symptom status, health status, fatigue). III. Evaluate the intermediate and long-term effects of these treatments on these patients and compare their impact on quality-of-life outcomes over 5 years.

OUTLINE: Quality-of-Life Assessment. Cancer Rehabilitation Evaluation System Short Form, CARES-SF; Symptom and Personal Information Questionnaire (including Symptom Distress Scale, MOS SF-36 Fatigue Scale, MOS SF-36 Health Perception Rating, Demographics); Cover Sheet.

PROJECTED ACCRUAL: Approximately 500 patients will be accrued over 7 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Patients must be eligible for and registered to SWOG-9133

PATIENT CHARACTERISTICS: Patients must be able to complete the questionnaires in English. If they are not able to complete questionnaires in English, patients may be registered to SWOG-9133 without participating in SWOG-9208.

The Symptom and Personal Information Questionnaire #1, the Cancer Rehabilitation Evaluation System Short Form (CARES-SF) and Cover Sheet must be completed prior to registration and randomization on SWOG-9133.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 263 (Actual)
Dates: Start 1994-04; Primary Completion 2003-09 (Actual); Study Completion 2005-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia A. Ganz, MD, Study Chair — Jonsson Comprehensive Cancer Center; Alice B. Kornblith, PhD, Study Chair — Dana-Farber Cancer Institute
Locations (11):
- United States (11):
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Beth Israel Medical Center, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee

REFERENCES:
- [Background] Ganz PA, Moinpour CM, McCoy S, et al.: Predictors of vitality (energy/fatigue) in early stage Hodgkin's disease (HD): results from Southwest Oncology Group (SWOG) study 9133. [Abstract] J Clin Oncol 22 (Suppl 14): A-6546, 569s, 2004.
- [Background] Ganz PA, Moinpour CM, Pauler DK, Kornblith AB, Gaynor ER, Balcerzak SP, Gatti GS, Erba HP, McCoy S, Press OW, Fisher RI. Health status and quality of life in patients with early-stage Hodgkin's disease treated on Southwest Oncology Group Study 9133. J Clin Oncol. 2003 Sep 15;21(18):3512-9. doi: 10.1200/JCO.2003.01.044. PMID 12972528
- [Derived] Moinpour CM, Unger JM, Ganz PA, Kornblith AB, Gaynor ER, Bowers MA, Gatti GS, Kaminski MS, Erba HP, Wang T, Yoon J, Press OW, Fisher RI. Seven-year follow-up for energy/vitality outcomes in early stage Hodgkin's disease patients treated with subtotal lymphoid irradiation versus chemotherapy plus radiation: SWOG S9133 and its QOL companion study, S9208. J Cancer Surviv. 2017 Feb;11(1):32-40. doi: 10.1007/s11764-016-0559-y. Epub 2016 Jul 12. PMID 27405732